CLINICAL TRIAL: NCT06822504
Title: ESPEN-EASO Sarcopenic Obesity (OS) Diagnostic Criteria Application in a COPD Cohort and OS Correlation to Diaphragmatic Thickness and Mobility for Determination of Tailored Pulmonary Rehabilitation Program: an Observational Study
Brief Title: Prevalence of Sarcopenic Obesity in COPD
Acronym: OS-BPCO
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Other Study IDs: 135/SR/24
Record Dates: First submitted 2024-06-07; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Sarcopenic Obesity; COPD
Keywords: sarcopenic obesity; COPD; diaphragmatic ultrasound
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Normal weight: 18.5< BMI > 24.99
- Overweight: 25< BMI > 29.99
- Obese: BMI > 30

SUMMARY:
The goal of this observational study is to the purpose is to apply of ESPEN/EASO criteria for the diagnosis of sarcopenic obesity and calculation of OS prevalence in a sample of COPD patients.

In addition, this study want to evaluate the impact of sarcopenic obesity on the respiratory function of COPD patients and the degree of severity of respiratory disease, assessed by spirometric examination; diaphragm thickness and excursion, by ultrasonographic study; performance, assessed by six-minute walk test (6-MWT); quality of life and degree of dyspnea (mMRC, Barthel dyspnea, S. George Respiratory Questionnaire); compliance and outcomes at the end of the respiratory rehabilitation course. Comparison with normal-weight patients with and without sarcopenia will help to better understand the clinical impact of sarcopenic obesity in this category of patients.

DETAILED DESCRIPTION:
From the review of the literature, there is a wide interest on both excess and deficient malnutrition in COPD patients, and more and more interest is being paid to sarcopenic obesity, which is a clinico-functional condition characterized by the coexisting presence of obesity, characterized by excess fat mass (FM), and sarcopenia, defined as reduced muscle mass and reduced function.

In the literature, there is no unambiguity on the diagnosis of sarcopenic obesity in terms of diagnostic criteria and cut-offs. Only recently, in 2022, have criteria for the diagnosis of sarcopenic obesity been defined through ESPEN/EASO consensus [Donini et al, 2022], shared by the international scientific community (Sarcopenic Obesity Global Leadership Initiative (SOGLI)).

The prevalence of sarcopenia in COPD patients is estimated to be 27% (He et al, 2023).Specifically, on the Italian population, at present it is known that the prevalence of sarcopenia in COPD is 24% (De Blasio et al, 2018), and that the prevalence of sarcopenia in obese individuals in the general population is 20 percent (Poggiogalle et al, 2026) but there are no recent studies showing what is the prevalence of sarcopenic obesity (diagnosed with ESPEN/EASO criteria) in COPD subjects in the Italian population.

This study aims to apply ESPEN/EASO criteria to identify obese sarcopenic patients and calculate the prevalence of sarcopenic obesity in COPD patients.

Finally, with this work, the investigators aim to study the impact of sarcopenic obesity on respiratory function (using both spirometric and ultrasonographic parameters to study the diaphragm), performance, degree of dyspnea, and thus quality of life in COPD patients, emphasizing the importance of early diagnosis in individuals with sarcopenic obesity in order to be able to intervene through targeted nutritional strategies to treat patients with chronic conditions, such as COPD, that significantly impact quality of life and health status.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 40 years of either sex;
* BMI >18.5
* COPD diagnosis according to the GOLD [2021 Global initiative for chronic obstructive lung disease] classification in the stable stage;
* Signing of informed consent after receiving all information about the study.

Exclusion Criteria:

* COPD not stabilized at the time of enrollment;
* BMI < 18.5
* presence of tracheostomy
* uncontrolled hypertension (systolic blood pressure > 160 mmHg, diastolic > 100 mmHg);
* hypotension (systolic blood pressure <100 mm Hg);
* Significant comorbidities that limit exercise tolerance;
* intercurrent infectious diseases, including HIV diagnosis;
* Patients diagnosed with malignancy in progress or in remission for less than 5 years;
* patients diagnosed with severe neurological, rheumatologic, or musculoskeletal diseases;
* patients with a history of thoracic surgery;
* presence of severe aortic stenosis, uncontrolled atrial/ventricular arrhythmia, recent cardiac ischemic event;
* cognitive impairment conditions that prevent full understanding of the study protocol (mental retardation, dementia, etc.) and/or adequate test performance compliance;
* failure to sign informed consent;
* any other serious medical condition that may interfere with data interpretation and safety or that may make the respiratory rehabilitation course difficult, limited, or uncomfortable.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable COPD admitted to the respiratory rehabilitation ward
Sampling Method: Non-Probability Sample
Enrollment: 236 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Diagnosis and calculation of sarcopenic obesity in COPD | From enrollment to the end of treatment at 4 weeks
  Application of ESPEN/EASO criteria for the diagnosis of sarcopenic obesity and calculation of OS prevalence in a sample of COPD patients.
  Sarcopenic obesity (ESPEN/EASO criteria): BMI &gt; 30 kg/m2 or CV (waist circumference) &gt; 102 cm M, 88 cm F E Clinical symptoms or clinical suspicion for OS screening or SARC-F ≥ 4 HGS + Sit-to-Stand test + BIA

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Roma, Roma, Italy